CLINICAL TRIAL: NCT07077018
Title: Fasting-Mimicking Diet as an Adjunct to Neoadjuvant Chemotherapy for Hormone-Receptor-Positive Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Kun Wang, Professor, Guangdong Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoFMD
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Fasting-Mimicking Diet; Breast Cancer; Neoadjuvant Chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FMD Group (Experimental)
  Interventions: Dietary Supplement: Fasting-mimicking diet (FMD) Group

INTERVENTIONS:
Dietary Supplement: Fasting-mimicking diet (FMD) Group — The FMD will consist of a triweekly 4-day regimen of a plant-based, calorie-restricted (827± 100 kcal on day 1；637 ± 100 kcal on days 2-4), low-carbohydrate, low-protein diet. The FMD will be repeated up to a maximum of eight consecutive cycles. Participants receive the FMD for 2 days prior to and on the day and one day after each cycle of chemotherapy.

SUMMARY:
This is a phase II, Single-Arm Clinical Study evaluating the efficacy and safety of a fasting-mimicking diet (FMD) combined with neoadjuvant chemotherapy in patients with ER-positive, HER2-negative breast cancer.

Participants will be assigned to Intervention group: 4-day FMD cycles (827± 100kcal/day on Day 1, 637± 100kcal/day on Days 2-4) synchronized with T-EC chemotherapy.

The primary endpoint is pathological complete response (pCR) rate. Secondary endpoints include metabolic changes, immune markers, quality of life, and safety (CTCAE v5.0). A total patients will be enrolled to detect a 15% pCR improvement (25% vs. 10%, α=0.05, power=80%).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ER-positive , HER2-negative invasive ductal carcinoma meeting at least one of the following:1)T1c-T2 N1 with histological grade 2 (ER 1-10%) or grade 3. 2)N2-N3 or grade 3 and/or Ki67 ≥40%. 3)T3-T4
* Age 18-75 years at enrollment
* Body mass index (BMI) ≥18.5 kg/m²
* Adequate hematological function:1）White blood cell count>3.0×10⁹/L.2)Absolute neutrophil count ≥1.5×10⁹/L.3)Platelets ≥100×10⁹/L.
* Adequate organ function:1）Total bilirubin ≤1.5 × upper limit of normal (ULN).2）ALT/AST ≤2.5 × ULN. 3）Alkaline phosphatase ≤5 × ULN.4）Creatinine clearance ≥50 mL/min-1)
* ECOG performance status 0-2
* Willing and able to provide written informed consent

Exclusion Criteria:

* Prior history of any malignancy (including contralateral breast cancer)
* Received any prior neoadjuvant chemotherapy cycle for current diagnosis
* Uncontrolled endocrine disorders:1)Diabetes mellitus requiring insulin or oral hypoglycemics.2)Hyper/hypothyroidism requiring medication
* Active autoimmune disease requiring systemic immunosuppressants
* Current use of antipsychotic medications
* Known hypersensitivity to FMD components (e.g., soy protein, milk protein, nuts)
* Pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-07-12 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | lmmediately after surgery
  The primary study endpoint of this trial was pCR, as defined as the absence of residual invasive disease on evaluation of surgical breast specimen and surgically-resected lymph nodes (i.e. ypT0/Tis ypN0）

CONTACTS AND LOCATIONS:
Overall Officials: Kun Wang, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, China